CLINICAL TRIAL: NCT01917331
Title: A Phase 3 Randomised Double Blind Randomised Parallel Multinational Trial Comparing a Fixed Combination of Beclometasone+Formoterol+Glycopyrrolate to Foster® in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Fixed Combination of Beclometasone + Formoterol + Glycopyrrolate Versus Foster® in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1207-PR-0091
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: spirometry; severe COPD; lung disease; fixed combination
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Beclomethasone; Formoterol Fumarate; Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beclometasone/Formoterol/Glycopyrrolate (Experimental): CHF 5993 pMDI 100/6/12.5 mcg 2 inhalations bid
  Interventions: Drug: Beclometasone/Formoterol/Glycopyrrolate
- Beclometasone/Formoterol (Active Comparator): Foster® 100/6 mcg 2 inhalations bid
  Interventions: Drug: Beclometasone/Formoterol

INTERVENTIONS:
Drug: Beclometasone/Formoterol/Glycopyrrolate — Active drug tested
  Other Names: BDP/FF/GB or CHF 5993 pMDI 100/6/12.5 mcg
  Arms: Beclometasone/Formoterol/Glycopyrrolate
Drug: Beclometasone/Formoterol — Active comparator
  Other Names: Foster® or CHF 1535 pMDI 100/6 mcg
  Arms: Beclometasone/Formoterol

SUMMARY:
Randomized,double-blind,multicenter,multinational,parallel-group,Phase III study to demonstrate the superiority of the triple fixed combination of Beclometasone+Formoterol+Glycopyrrolate (BDP/FF/GB) administered via pMDI over the equivalent dose of Foster® in COPD (Chronic Obstructive Pulmonary Disease) patients after 52 weeks of treatment

DETAILED DESCRIPTION:
This 52-week randomised 2 parallel groups study aimed at evaluating the superiority of fixed triple therapy with ICS/LABA/LAMA compared to ICS/LABA in severe to very severe COPD patients.

Patients' eligibility was checked during the screening visit including the review of medical history, spirometry assessments, routine labs, physical examination, 12-lead ECG, vital signs measurement. This visit was followed by a 2-week open-label run-in period under Foster® (BDP/FF 400/24 µg total daily dose). Eligible patients were then randomised to either fixed triple therapy BDP/FF/GB or BDP/FF. During the 52-week treatment period, completing patients did have 5 subsequent visits post randomisation scheduled respectively after 4 (Visit 3), 12 (Visit 4), 26 (Visit 5), 40 (Visit 6) and 52 (Visit 7) weeks of treatment.

During these, pre-dose and post-dose spirometry, 12-lead ECG, vital signs, dyspnea assessments were performed. Rescue medication use, compliance with the treatment and EXACT-PRO questionnaire were recorded daily (via an electronic diary) during the run-in and randomised treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 40 years with a diagnosis of COPD
* Current smokers or ex-smokers
* A post-bronchodilator FEV1 < 50% of the predicted normal value and a post- bronchodilator FEV1/FVC < 0.7
* At least one exacerbation in the 12 months preceding the screening visit

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of asthma or history of allergic rhinitis or atopy
* Patients treated with non-cardioselective β-blockers in the month preceding the screening visit
* Patients treated for exacerbations in the 4 weeks prior to screening visit
* Patients treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study or if taken as PRN
* Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia
* Known respiratory disorders other than COPD
* Patients who have clinically significant cardiovascular condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1368 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pre-dose and 2-hour post-dose morning FEV1 at week 26 and TDI score at week 26 | week 26
  * Change from baseline in pre-dose morning FEV1 at Week 26.
  * Change from baseline to the 2-hour post-dose value of FEV1 at Week 26.
  * TDI focal score at Week 26

SECONDARY OUTCOMES:
COPD exacerbation rate | week 52
  Moderate and severe COPD exacerbation rate over 52 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dave SINGH, MD, Principal Investigator — University Hospital of South Manchester, MANCHESTER M23 9 QZ, UK
Locations (1):
- Dr Beatrix BALINT, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanfleteren L, Fabbri LM, Papi A, Petruzzelli S, Celli B. Triple therapy (ICS/LABA/LAMA) in COPD: time for a reappraisal. Int J Chron Obstruct Pulmon Dis. 2018 Dec 12;13:3971-3981. doi: 10.2147/COPD.S185975. eCollection 2018. PMID 30587953
- [Background] Singh D, Fabbri LM, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy delays COPD clinically important deterioration vs ICS/LABA, LAMA, or LABA/LAMA. Int J Chron Obstruct Pulmon Dis. 2019 Feb 28;14:531-546. doi: 10.2147/COPD.S196383. eCollection 2019. PMID 30880943
- [Background] Singh D, Fabbri LM, Corradi M, Georges G, Guasconi A, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy in patients with symptomatic COPD and history of one moderate exacerbation. Eur Respir J. 2019 May 18;53(5):1900235. doi: 10.1183/13993003.00235-2019. Print 2019 May. PMID 30792343
- [Result] Singh D, Papi A, Corradi M, Pavlisova I, Montagna I, Francisco C, Cohuet G, Vezzoli S, Scuri M, Vestbo J. Single inhaler triple therapy versus inhaled corticosteroid plus long-acting beta2-agonist therapy for chronic obstructive pulmonary disease (TRILOGY): a double-blind, parallel group, randomised controlled trial. Lancet. 2016 Sep 3;388(10048):963-73. doi: 10.1016/S0140-6736(16)31354-X. Epub 2016 Sep 1. PMID 27598678
- See also: EU Clinical Trial Register - Study Record including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CCD-1207-PR-0091
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1207-PR-0091.pdf